CLINICAL TRIAL: NCT07179354
Title: Comparative Assessment of Three-Dimensional Soft and Hard Tissue Changes Following Rapid Maxillary Expansion With Face Mask, Mini Maxillary Protractor, and Modified Splints, Elastics, and Chin Cup Protocols in Patients With Class III Malocclusion: A Prospective Randomized Controlled Clinical Trial
Brief Title: Comparative 3D Assessment of Class III Malocclusion Treatments
Acronym: CLASSIII-3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gokhan Coban, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024\44
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Class III Skeletal Malocclusion
Keywords: Class III malocclusion; RME/FM; Mini maxillary protractor; SEC III; 3D stereophotogrammetry; Soft tissue; Cephalometry
MeSH Terms: conditions — Malocclusion, Angle Class III | interventions — Masks

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design, where participants with Class III skeletal malocclusion are randomly assigned to one of three treatment groups: rapid maxillary expansion with face mask (RME/FM), mini maxillary protractor (MMP), or modified splints with elastics and chin cup (SEC III). Additionally, a control group consisting of untreated patients with similar malocclusion characteristics from archival records is included for comparison. Each treatment group receives its specific intervention simultaneously, and outcomes are compared among all groups to evaluate the efficacy of each protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RME/FM Group (Rapid Maxillary Expansion with Face Mask) (Experimental): Participants in this group received rapid maxillary expansion using a bonded expander, followed by protraction with a face mask. This protocol aims to advance the maxilla in patients with Class III skeletal malocclusion.
  Interventions: Device: Rapid Maxillary Expansion with Face Mask (RME/FM)
- MMP Group (Mini Maxillary Protractor) (Experimental): This group was treated with the Mini Maxillary Protractor (MMP), a custom-designed intraoral appliance used to achieve orthopedic maxillary protraction without external devices. The aim is to promote maxillary advancement in growing Class III patients.
  Interventions: Device: Mini Maxillary Protractor (MMP)
- Modified SEC III Group (Modified Splints with Elastics and Chin Cup) (Experimental): Participants in this group were treated using modified splints with intermaxillary elastics and a chin cup (SEC III protocol). The protocol is designed to restrict mandibular growth and enhance maxillary positioning in patients with skeletal Class III malocclusion.
  Interventions: Device: Modified Splint with Elastics and Chin Cup (Modified SEC III)
- Control Group (Untreated group selected from archival records) (No Intervention): This group includes untreated patients with Class III skeletal malocclusion, selected from archival records. No intervention was administered. The group serves as a baseline comparison for evaluating treatment effects.

INTERVENTIONS:
Device: Rapid Maxillary Expansion with Face Mask (RME/FM) — A tooth- and tissue-borne rapid maxillary expansion appliance with an expansion screw was used to achieve transverse maxillary expansion, followed by Petit-type face mask therapy. Expansion protocol: two quarter-turns per day for 10-14 days, then one quarter-turn per day until cusp-to-cusp relationship was achieved. Face mask elastics applied 16 hours/day at 350-500 g per side, with a 30° downward and forward vector relative to the occlusal plane.
  Arms: RME/FM Group (Rapid Maxillary Expansion with Face Mask)
Device: Mini Maxillary Protractor (MMP) — An intraoral mini maxillary protraction appliance was used to advance the maxilla. Force was applied through intraoral elastics connected to intraoral anchorage units. The protocol was designed to deliver orthopedic forward traction of the maxilla without an external face mask.
  Arms: MMP Group (Mini Maxillary Protractor)
Device: Modified Splint with Elastics and Chin Cup (Modified SEC III) — A modified splint appliance combined with intraoral elastics and an orthopedic chin cup was used to achieve skeletal mandibular retrusion and Class III correction. The appliance applied orthopedic forces through combined vertical and horizontal components, promoting backward positioning of the mandible while maintaining transverse maxillary relationships.
  Arms: Modified SEC III Group (Modified Splints with Elastics and Chin Cup)

SUMMARY:
This clinical trial compares three different treatment methods used to correct jaw problems in children with Class III malocclusion (a condition where the lower jaw is positioned forward relative to the upper jaw). The treatments include:

Rapid maxillary expansion with face mask (RME/FM),

Mini maxillary protractor (MMP),

Modified splints with elastics and chin cup (SEC III).

The study aims to understand how each treatment affects the bones and soft tissues of the face, such as how much the upper jaw moves forward or the lower jaw moves backward, as well as changes in teeth alignment and facial appearance. Results showed that different treatments work best for different aspects: some are better for moving the upper jaw forward, while others are better for repositioning the lower jaw. This information helps doctors choose the most suitable treatment plan for each patient.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical trial evaluates and compares the skeletal and three-dimensional soft tissue effects of three orthopedic treatment protocols in growing patients with Class III skeletal malocclusion. A total of 43 patients were randomly assigned to one of three treatment groups: rapid maxillary expansion with face mask (RME/FM), mini maxillary protractor (MMP), and modified splints with elastics and chin cup (SEC III). Additionally, a control group was formed from archival records of untreated patients with similar malocclusion characteristics.

Patients underwent comprehensive evaluation before and after treatment, including lateral cephalometric radiographs and 3D stereophotogrammetry to capture skeletal and soft tissue changes. Key parameters measured were maxillary and mandibular skeletal movements, dental inclination changes, overjet and overbite adjustments, as well as facial soft tissue displacement and angular measurements.

The study's design ensured rigorous randomization and controlled conditions to objectively assess the efficacy of each treatment protocol. The outcomes provide insight into how each method influences skeletal advancement or retrusion, dental positioning, and facial profile alterations, offering guidance for personalized treatment planning in orthodontic practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have not completed their growth spurt (9-12 years old)
* Overjet ≤ 0 mm (patients with negative overjet must be De Nevreze positive)
* ANB ≤ 0°, Witts < 1
* Good oral hygiene and healthy periodontal tissues
* SN-GoGn angle between 26° and 38°
* No congenital or acquired tooth loss (excluding third molars)
* Body mass index (BMI) between 18-26 kg/m²
* No systemic, local, or endocrinological diseases

Exclusion Criteria:

* Presence of any syndrome or developmental deformity
* Previous orthodontic treatment
* Allergy to any metal or acrylic
* Presence of any systemic disease affecting treatment
* SN-GoGn angle > 38°
* Presence of temporomandibular joint disorders

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Three-dimensional changes in soft tissues | baseline to post-treatment (≈ 9 months)
  3D stereophotogrammetry used to assess overall soft tissue profile changes, including facial convexity and lip-chin parameters.

SECONDARY OUTCOMES:
Two dimensional changes in skeletal parameters of the maxilla and mandible | Baseline (pre-treatment) to post-treatment (≈ 9 months)
  Lateral cephalometric radiographs used to evaluate overall skeletal changes in maxillary and mandibular positions, as well as dental parameters including overjet and overbite.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Çoban, Associate Professor, PhD,, Principal Investigator — Erciyes University, Faculty of Dentistry, Department of Orhodontics; Tuba Ünlü Çiftçi, Research Assistant, Principal Investigator — Erciyes University, Faculty of Dentistry, Department of Orhodontics
Locations (1):
- Erciyes University, Faculty of Dentistry, Department of Orthodontics, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset is limited to a small number of pediatric patients and was collected solely for internal academic research purposes.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT07179354/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT07179354/ICF_001.pdf